CLINICAL TRIAL: NCT05856487
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of NVP-2203 Tablet in Patients
Brief Title: To Evaluate the Safety and Efficacy of NVP-2203 Tablet in Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVP-2203_P3
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NVP-2203 (Experimental): NVP-2203 Plus other Placebo for up to 8 weeks, oral dose
  Interventions: Drug: NVP-2203; Drug: NVP-2203-R1 Placebo; Drug: NVP-2203-R2 Placebo; Drug: NVP-2203-R3 Placebo
- NVP-2203-R1 (Active Comparator): NVP-2203-R1 Plus other Placebo for up to 8 weeks, oral dose
  Interventions: Drug: NVP-2203-R1; Drug: NVP-2203 Placebo; Drug: NVP-2203-R2 Placebo
- NVP-2203-R2 (Active Comparator): NVP-2203-R2 Plus other Placebo for up to 8 weeks, oral dose
  Interventions: Drug: NVP-2203-R2; Drug: NVP-2203 Placebo; Drug: NVP-2203-R1 Placebo; Drug: NVP-2203-R3 Placebo
- NVP-2203-R3 (Active Comparator): NVP-2203-R3 Plus other Placebo for up to 8 weeks, oral dose
  Interventions: Drug: NVP-2203-R3; Drug: NVP-2203 Placebo; Drug: NVP-2203-R1 Placebo; Drug: NVP-2203-R2 Placebo

INTERVENTIONS:
Drug: NVP-2203 — Take it once daily for 8 weeks orally.
  Arms: NVP-2203
Drug: NVP-2203-R1 — Take it once daily for 8 weeks orally.
  Arms: NVP-2203-R1
Drug: NVP-2203-R2 — Take it once daily for 8 weeks orally.
  Arms: NVP-2203-R2
Drug: NVP-2203-R3 — Take it once daily for 8 weeks orally.
  Arms: NVP-2203-R3
Drug: NVP-2203 Placebo — Take it once daily for 8 weeks orally.
  Arms: NVP-2203-R1; NVP-2203-R2; NVP-2203-R3
Drug: NVP-2203-R1 Placebo — Take it once daily for 8 weeks orally.
  Arms: NVP-2203; NVP-2203-R2; NVP-2203-R3
Drug: NVP-2203-R2 Placebo — Take it once daily for 8 weeks orally.
  Arms: NVP-2203; NVP-2203-R1; NVP-2203-R3
Drug: NVP-2203-R3 Placebo — Take it once daily for 8 weeks orally.
  Arms: NVP-2203; NVP-2203-R2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety NVP-2203 in patients

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, parallel-group, phase 3 clinical trial to evaluate efficacy and safety of NVP-2203 in patients

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 19 years of age
* Primary hypercholesterolemia
* Subjects who have ability to comprehend the contents of study and before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* The subject not meet the specified LDL-C level
* Patients who were diagnosed with a malignant tumor within five years before Visit
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
% change in LDL-C level from baseline | Week 8
  change in LDL-C level

SECONDARY OUTCOMES:
% change in lipid panel from baseline | Week 4, 8
  change in lipid panel

CONTACTS AND LOCATIONS:
Overall Officials: SH Lee, MD, Principal Investigator — Severance Hospital
Locations (1):
- NVPhealthcare, Suwon, Gyeonggi-do, South Korea